CLINICAL TRIAL: NCT06049810
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Randomized Withdrawal and Retreatment Phase III Clinical Trial Evaluating the Efficacy and Safety of Subcutaneous Injection of IBI112 in the Treatment of Moderate to Severe Plaque Psoriasis.
Brief Title: IBI112 in Moderate to Severe Plaque Psoriasis With Randomized Withdrawal and Re-treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI112A302CN
Record Dates: First submitted 2023-09-13; First posted 2023-09-22 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 3 (Experimental): Participants receive Dose 1 IBI112 through week 8 & Dose 2 IBI112 on week 20 & Dose 1 IBI112 through week 44
  Interventions: Drug: IBI112
- Group 4 (Experimental): Participants receive Dose 1 IBI112 through week 8 & Dose 3 IBI112 through week 44
  Interventions: Drug: IBI112
- Group 6 (Experimental): Participants receive Dose 1 IBI112 through week 8 & Dose 3 IBI112 on week 20 & Dose 1 IBI112 through week 44
  Interventions: Drug: IBI112
- Group 5 (Placebo Comparator): Participants receive Dose 1 IBI112 through week 8 & Dose 3 IBI112 on week 20 & placebo through week 44
  Interventions: Drug: IBI112/placebo
- Group 1 (Experimental): Participants receive Dose 1 IBI112 through week 8 & Dose 2 IBI112 through week 44
  Interventions: Drug: IBI112
- Group 2 (Placebo Comparator): Participants receive Dose 1 IBI112 through week 8 & Dose 2 IBI112 on week 20 & placebo through week 44
  Interventions: Drug: IBI112/placebo

INTERVENTIONS:
Drug: IBI112 — Participants receive Dose 1 IBI112 through week 8 & Dose 2 IBI112 on week 20 & Dose 1 IBI112 through week 44
  Arms: Group 3
Drug: IBI112/placebo — Participants receive Dose 1 IBI112 through week 8 & Dose 2 IBI112 on week 20 & placebo through week 44 by subcutaneous injection
  Arms: Group 2
Drug: IBI112/placebo — Participants receive Dose 1 IBI112 through week 8 & Dose 3 IBI112 on week 20 & placebo through week 44
  Arms: Group 5
Drug: IBI112 — Participants receive Dose 1 IBI112 through week 8 & Dose 3 IBI112 on week 20 & Dose 1 IBI112 through week 44
  Arms: Group 6
Drug: IBI112 — Participants receive Dose 1 IBI112 through week 8 & Dose 3 IBI112 through week 44
  Arms: Group 4
Drug: IBI112 — Participants receive Dose 1 IBI112 through week 8 & Dose 2 IBI112 through week 44 by subcutaneous injection
  Arms: Group 1

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of IBI112 in the treatment of participants with moderate to severe psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of plaque-type psoriasis for at least 6 months;
2. Psoriasis Area and Severity Index (PASI) score of 12 or greater, AND static Physician's Global Assessment (sPGA) score of 3 (moderate) or greater; Psoriasis covering at least 10% of body surface area;
3. Must be a candidate for either systemic therapy or phototherapy for psoriasis.

Exclusion Criteria:

1. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (for example, compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments
2. Participants who have ever received IBI112 or IL-23 inhibitor
3. History or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
4. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest of the participant
5. Is pregnant, nursing, or planning a pregnancy (both men and women) within 6 months following the last administration of the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a Psoriasis Area and Severity Index (PASI) 90 Response | Week 56

SECONDARY OUTCOMES:
Percentage of participants with a PASI75 Response | Week 56
Percentage of participants with a PASI100 Response | Week 56
Percentage of participants with a static Investigator's Global Assessment (sIGA) score of 0 or 1 | Week 56
Percentage of participants with Dermatology Life Quality Index (DLQI) Score | Week 56
Percentage of participants with a sIGA score of 0 | Week 56
Cumulative Maintenance Rate of PASI 90 Response Through Week 56 to Evaluate Loss of a PASI 90 Response | Week 56
Changes of PASI Scores participants who relapse and retreatment | Week 56
Changes of sIGA score in participants who relapse and retreatment | Week 56

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No